CLINICAL TRIAL: NCT04667702
Title: HPV Vaccine Hesitancy Among Indiana Youth With Cancer and Blood Diseases
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Scott L Coven, DO, MPH, Assistant Professor of Pediatrics, Indiana University
Other Study IDs: 2010192007
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Human Papilloma Virus Vaccine Hesitancy
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient Focused Interviews
  Interventions: Behavioral: Interviews
- Caregiver Focused Interviews
  Interventions: Behavioral: Interviews
- Healthcare Provider Focused Interviews
  Interventions: Behavioral: Interviews

INTERVENTIONS:
Behavioral: Interviews — We will conduct a phone or virtual interview with patients with sickle cell disease or cancer, caregivers and their healthcare providers.

SUMMARY:
For the identified groups of patients (survivors of childhood cancer and youth with sickle cell disease) the investigators want to better understand the barriers to, and facilitators of, HPV vaccination. Through HCP interviews the investigators will also assess both attitudinal and logistical obstacles to HPV vaccination. Some subspecialty HCPs may believe, for instance, that it is the primary care provider's responsibility to vaccinate or they may be unfamiliar with the requirement to enter vaccination data into CHIRP. Also, in some cases HPV vaccine may not be readily available in subspecialty clinic locations and/or subspecialty HCPs may not be Vaccines for Children (VFC) providers. Participants: the investigators will focus on two patient groups: survivors of childhood cancer, which includes children aged 9-21 years who have completed active therapy for cancer and are eligible for vaccination, and sickle cell disease, which includes children aged 9-21 years with a diagnosis of sickle cell disease. The investigators will recruit parents of children aged 9-21 years and older adolescents aged 18-21 years. For pediatric patients, the investigators selected a lower age of 9 years because HPV vaccine is licensed down to 9 years of age, and an upper limit of 21 years, as that is considered the upper bound of adolescence by the American Academy of Pediatrics. For patients 9-17 years of age, only parents will be interviewed by video or phone because parents are the vaccine decision-makers. For patients 18-21 years of age, the investigators will interview both young adults and their parents, because, while the young adult has legal decision-making capacity, in reality, the decision is frequently made jointly by the young adult and parent, and older adolescents are frequently unwilling to go against their parents' wishes. All research procedures will be conducted in English. Participants will be excluded if they have an intellectual disability or severe medical illness such that they are unable to consent or to understand the questions.

ELIGIBILITY:
Inclusion Criteria:

* Age 9-21 years of age for patients with sickle cell disease or cancer.
* Caregiver of patient with sickle cell disease or cancer.
* Healthcare provider of patient with sickle cell disease or cancer.

Exclusion Criteria:

* n/a

Ages: 9 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with sickle cell disease or cancer. Caregivers of patients with sickle cell disease or cancer. Healthcare providers of patients with sickle cell disease or cancer.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Vaccine Hesitancy 5 point Likert scale | 1 Day
  Patients will be scored using scale: 1=strongly disagree; 2=disagree; 3=neither agree nor disagree; 4=agree; and 5=strongly agree; lower scores mean less confidence/more hesitancy; higher scores mean more confidence/less hesitancy.
Vaccine Hesitancy 5 point Likert scale | 1 Day
  Caregivers will be scored using scale: 1=strongly disagree; 2=disagree; 3=neither agree nor disagree; 4=agree; and 5=strongly agree; lower scores mean less confidence/more hesitancy; higher scores mean more confidence/less hesitancy.
Hesitancy or Confidence of counseling or giving the HPV vaccine of health care providers | 1 Day
  Interview Results - no scale available. Themes and descriptive.

CONTACTS AND LOCATIONS:
Locations (1):
- Riley Hospital for Children - Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No